CLINICAL TRIAL: NCT05446480
Title: Potential Off-label Use of Desloratadine to Mitigate Inflammation Caused by PPE-induced Heat Stress
Brief Title: Role of Desloratadine in Reducing Inflammation From Occupational Heat Strain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Victoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21-0616
Record Dates: First submitted 2022-06-13; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-05

CONDITIONS: Heat Stress, Exertional; Inflammatory Response; Firefighter Personal Protective Equipment
MeSH Terms: conditions — Heat Stress Disorders | interventions — desloratadine

STUDY DESIGN:
Intervention Model Description: Own-control study - all participants perform each trial arm/intervention separated by a washout period. Order of trials is randomized for each participant.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Desloratadine (Experimental): Desloratadine (Aerius) 10mg compounded to oral pill
  Interventions: Drug: Desloratadine
- Inert Placebo (Experimental): Placebo 10mg compounded to oral pill
  Interventions: Drug: Placebo
- No Intervention (Experimental): No intervention: neither drug nor placebo
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Desloratadine — Oral ingestion 10mg pill 2 hours prior to heat strain trial. Second 10mg dose 24-hours later.
  Other Names: Desloratadine (Aerius)
  Arms: Desloratadine
Drug: Placebo — Oral ingestion 10mg inert pill 2 hours prior to heat strain trial. Second dose 24-hours later.
  Other Names: Inert Placebo
  Arms: Inert Placebo
Other: No Intervention — No pill ingestion during the trial - to discern the presence of a placebo effect from baseline inflammatory response
  Other Names: Neither Drug nor Placebo
  Arms: No Intervention

SUMMARY:
The aim of this initial investigational study is to compare the effect of desloratadine on the inflammatory responses to heat stress in firefighters exercising in their personal protective equipment.

DETAILED DESCRIPTION:
Significant heat strain where temperatures approach and exceed 39.0 degrees celsius is known to increase intestinal permeability and induce a graded systemic inflammatory response which includes increases in interleukin-6, tumor necrosis factor alpha, and c-reactive protein. Recent data examining firefighters found fire service instructors possessed greater resting levels of inflammatory markers and that 18-29% of the variation in these markers could be explained by frequency of heat strain. Firefighters themselves are susceptible to core temperatures ranging between 38.5 and 39.0C in as little as 2-3 work cycles. Considering resource limitation in the fire service, such workloads is a realistic possibility when at structural fires, particularly for first alarm apparatus.

Though there is a well-defined role of the inflammatory response in adaptive changes, elevated resting levels begs the question of whether such frequency of exposure and acute inflammatory flux in fire service workers may contribute to chronic elevations of inflammatory markers and altered disease risk. Elevations in c-reactive protein are associated with cardiovascular risk with studies indicating a causative role of monomeric c-reactive protein in platelet activation and thrombus growth.

Cooling methods save for cryotherapy have demonstrated limited to mild effectiveness for mitigating the inflammatory responses to heat strain resulting in no solution to attenuate acute inflammatory responses. The mast-cell stabilizing properties of desloratadine and its safety profile make it an interesting candidate for investigating its use in this context.

This study seeks to determine whether 10mg desloratadine taken before and 24h after exertional heat strain to a core temperature to a core temperature of 39.5 degrees celsius reduces the associated inflammatory response measured over a 72-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated willingness to participate in the study and adhere to procedures by signing a written informed consent
* Biological males aged 19-50
* Successful Physical Activity Readiness Questionnaire (PAR-Q)
* Ability to swallow core temperature capsule
* VO2Max >35 mL/kg/min
* No allergy or current dosage of H1 histamine receptor antagonists
* Participants must be in good health with no 'Category A' diseases/conditions outlined in National Fire Protection Association (NFPA) 1582 (https://www.iafc.org/docs/default-source/1vcos/vws_rrkit_nfpa-1582.pdf?sfvrsn=ca9b9f0d_2)

Exclusion Criteria:

* Biological females
* Males below age of 19, and 51-years or older
* Unsuccessful PAR-Q
* VO2Max below 35 mL/kg/min
* Allergy to H1 histamine receptor antagonists
* Esophageal constriction (inability to swallow core temperature capsule)
* Any condition or disease listed as 'Category A' in NFPA 1582 that would disqualify a person as a firefighter.
* Current use of NSAIDS or steroid drugs (oral or nasal).
* Consumption of caffeine, nicotine, or alcohol in the preceding 12-hours.
* Dehydration (urine specific gravity over 1.030)
* Recent cold/flu (at least 7-days clear of symptom resolution)
* No use of antibiotics in preceding 14-days.
* Dosing of medication that is known to exhibit adverse reactions with desloratadine dosing.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change in serum cortisol | Before, immediately following, and 2-hours following exertional heat strain
  Assessment of changes in serum cortisol within and between interventions measured via venipuncture and ELISA
Change in serum interleukin-6 and ELISA | Before, immediately following, and 2-hours following exertional heat strain
  Assessment of changes in serum interleukin-6 within and between interventions measured via venipuncture and ELISA
Change in serum c-reactive protein | Before, immediately following, and 24, 48, and 72-hours following exertional heat strain
  Assessment of changes in serum c-reactive protein within and between interventions measured via venipuncture and ELISA
Change in serum tumor necrosis factor alpha | Before, immediately following, and 2-hours following exertional heat strain
  Assessment of changes in serum tumor necrosis factor alpha within and between interventions measured via venipuncture and ELISA.

SECONDARY OUTCOMES:
Change in body mass | Before and immediately after exertional heat strain
  Trial arm differences in fluid loss estimated via differences between before-after body mass.
Differences in core body heat storage | Before and immediately after exertional heat strain
  Trial arm differences in the change in core body temperature during heating.

OTHER OUTCOMES:
Differences in Cerebral Blood Flow | Before and immediately after (following assessment of outcome 8 and 9) exertional heat strain
  Within and between intervention differences in cerebral blood flow changes via vascular duplex ultrasound and hypercapnia
Differences in heart rate (HR) and heart rate variability (HRV) | Before and immediately after exertional heat strain
  Within and between intervention differences in HR and HRV
Differences in brain blood oxygenation of prefrontal cortex | Before and immediately after exertional heat strain
  Within and between intervention differences in prefrontal cortex oxygenation via near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Lynneth Stuart-Hill, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data, if used in a publication, may be available in a data repository with all identifiers removed.